CLINICAL TRIAL: NCT00732082
Title: Phase I Study of Soluble LAG-3 (IMP321) and Gemcitabine in Patients With Advanced Pancreas Cancer
Brief Title: Lag-3 and Gemcitabine for Treatment of Advanced Pancreas Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company manufacturing study drug was unable to continue production.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0265
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Pancreatic Neoplasms
Keywords: LAG-3 and gemcitabine treatment for advanced pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose Level 0 (Active Comparator): Gemcitabine (1 mg/m2 over 30 min) will be given on days 1, 8, and 15 of a 28 day cycle.
  Interventions: Drug: Gemcitabine
- Dose Level 1 (Experimental): Gemcitabine (1 mg/m2 over 30 min) will be given on days 1, 8, and 15 of a 28 day cycle.
  IMP321 3 mg SQ anterior surface of either the right or left thigh on Day 2.
  The subsequent doses will be given by subcutaneous injection on the contralateral thigh.
  Each single injection will be separated by a 13-day administration free period.
  Interventions: Drug: Gemcitabine; Biological: LAG-3
- Dose Level 2 (Experimental): Gemcitabine (1 mg/m2 over 30 min) will be given on days 1, 8, and 15 of a 28 day cycle.
  IMP321 6.5 mg SQ anterior surface of either the right or left thigh on Day 2.
  The subsequent doses will be given by subcutaneous injection on the contralateral thigh.
  Each single injection will be separated by a 13-day administration free perio
  Interventions: Drug: Gemcitabine; Biological: LAG-3
- Dose Level 3 (Experimental): Gemcitabine (1 mg/m2 over 30 min) will be given on days 1, 8, and 15 of a 28 day cycle.
  IMP321 13 mg SQ anterior surface of either the right or left thigh on Day 2.
  The subsequent doses will be given by subcutaneous injection on the contralateral thigh.
  Each single injection will be separated by a 13-day administration free perio
  Interventions: Drug: Gemcitabine; Biological: LAG-3
- Dose Level 4 (Experimental): Gemcitabine (1 mg/m2 over 30 min) will be given on days 1, 8, and 15 of a 28 day cycle.
  IMP321 26 mg SQ anterior surface of either the right or left thigh on Day 2.
  The subsequent doses will be given by subcutaneous injection on the contralateral thigh.
  Each single injection will be separated by a 13-day administration free perio
  Interventions: Drug: Gemcitabine; Biological: LAG-3

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Biological: LAG-3
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4

SUMMARY:
The overall purpose of this research is to evaluate the safety and toxicity of an investigational medication, IMP321, in patients being treated with gemcitabine. IMP321 is a synthetic protein (made in the laboratory to simulate a protein that your body makes on its own) and was designed to stimulate the immune system with the overall objective of improving the body's capacity to react to your pancreas cancer.

DETAILED DESCRIPTION:
This is a phase I, single center, open label, non-randomized, dose-escalation phase I study performed in the ambulatory setting in patients receiving first line chemotherapy for unresectable pancreas cancer with gemcitabine weekly and the investigational agent IMP321. IMP321 will be given at D2 and D16 of a 4-week cycle, for a period of 6 months. The hypothesis of this study is that IMP321 is safe for human administration. Additionally we hypothesize that IMP321 elicits an immunomodulatory effect that is therapeutic in the treatment of pancreas cancer.

Primary Objectives

* To evaluate the safety and tolerability of repeated IMP321 subcutaneous injections in patients being treated with gemcitabine for advanced pancreas cancer.
* To determine any dose limiting toxicities of IMP321 in patients being treated with gemcitabine for advanced pancreas cancer.

Secondary Objectives

* To describe the pharmacokinetics of the last IMP321 subcutaneous injection compared to the first one, in a limited number of patients.
* To determine the pharmacodynamics of IMP321 therapy by:
* Quantify peripheral blood Treg (CD4+CD25+FoxP3+ T cells) in pancreatic cancer patients before and during treatment with IMP321 by flow cytometry.
* Evaluate the B- and T-cell responses to the pancreatic cancer-expressed antigen, mesothelin, by testing for antibodies and T-cell response by ELISpot.
* To evaluate the clinical response and time to disease progression with computed tomography examinations at two month intervals (current standard of care in gemcitabine-treated patients).

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a newly diagnosed, histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma (primary tumor or metastasis). The histological slides or blocks must be available for review.
* Patient must have advanced disease (characterized by metastasis or locally advanced disease), or unable to undergo surgical treatment due to extent of disease or pre-existing health conditions precluding surgical treatment.
* Measurable or evaluable disease: RECIST Criteria will be used to assess and survey extent of disease
* Patients must be ≥ 18 years old.
* Performance Status: Karnofsky Performance Status (KPS) ≥ 70
* Life Expectancy > 12 weeks.
* No previous history of chemotherapy for pancreas cancer in the metastatic setting prior to the start of protocol treatment.
* Patients must have recovered from uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Patients must have adequate bone marrow function defined as an absolute neutrophil count >1,500/mm3, platelet count >100,000/mm3 and hemoglobin >10 g/dl.
* Patients must have adequate renal function defined as serum creatinine ≤ 2.0 mg/dl or creatinine clearance ≥ 60 ml/min/1.73m2 for patients with creatinine levels above 2.0 mg/dl.
* Patients must have adequate hepatic function with total bilirubin ≤ 1.5 times the institutional normal value and AST ≤ 2 times the institutional normal value.
* Patient must have no prior or current active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, systemic vasculitis, scleroderma, psoriasis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, sarcoidosis or other rheumatologic disease. Asthma and chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable.
* The patient with previous history of malignancy is eligible for this study only if the patient meets the following criteria for cancer survivor:

  * (i) patient has undergone potentially curative therapy for all prior malignancies;
  * (ii) patient has been considered disease free for at least 5 years.
* For all sexually active patients, the use of adequate barrier contraception (hormonal or barrier method of birth control) will be required during therapy, prior to study entry and for the duration of study participation. Patients must agree to refrain from becoming pregnant 2 years after beginning treatment with IMP321. Non-pregnant status will be determined in all women of childbearing potential.
* After being informed of the treatment involved, patients must give written consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.

Exclusion Criteria:

* Patient is currently receiving other investigational agents.
* Pregnant and nursing women patients are not eligible.
* Patients known to be HIV (patient self-report) positive are ineligible because of the potential inability to modulate immune responses.
* Patients with a QTc of >460 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of repeated IMP321 subcutaneous injections in patients being treated with gemcitabine for advanced pancreas cancer. | 6 months
To determine the dose limiting toxicities of IMP321 in patients being treated with gemcitabine for advanced pancreas cancer. | 6 months

SECONDARY OUTCOMES:
To describe the pharmacokinetics of the last IMP321 subcutaneous injection compared to the first one, in a limited number of patients. | Pre-dose, 2 hours, 4 hours, 8 hours, 24 hours, 72 hours, and 96 hours after IMP321 administration
  Performed only in patients enrolled in dose level 3 and 4.
To determine the pharmacodynamics of IMP321 therapy | 6 months
  1. Quantify peripheral blood Treg (CD4+ CD25+ Fox P3+ Tcells) in pancreatic cancer patients before and during treatment with IMP321 by flow cytometry.
  2. Evaluate the B- and T-cell responses to the pancreatic cancer-expressed antigen, mesothelin, by testing for antibodies and T-cell response by ELISpot
To evaluate the clinical response and time to disease progression with computed tomography examinations at two month intervals (current standard of care in gemcitabine-treated patients). | survival

CONTACTS AND LOCATIONS:
Overall Officials: William G. Hawkins, M.D., Principal Investigator — Washington Univerisity
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Storniolo AM, Allerheiligen SR, Pearce HL. Preclinical, pharmacologic, and phase I studies of gemcitabine. Semin Oncol. 1997 Apr;24(2 Suppl 7):S7-2-S7-7. PMID 9194473
- [Background] Green MR. Gemcitabine safety overview. Semin Oncol. 1996 Oct;23(5 Suppl 10):32-5. PMID 8893879
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Linehan DC, Goedegebuure PS. CD25+ CD4+ regulatory T-cells in cancer. Immunol Res. 2005;32(1-3):155-68. doi: 10.1385/IR:32:1-3:155. PMID 16106066
- [Background] Liyanage UK, Moore TT, Joo HG, Tanaka Y, Herrmann V, Doherty G, Drebin JA, Strasberg SM, Eberlein TJ, Goedegebuure PS, Linehan DC. Prevalence of regulatory T cells is increased in peripheral blood and tumor microenvironment of patients with pancreas or breast adenocarcinoma. J Immunol. 2002 Sep 1;169(5):2756-61. doi: 10.4049/jimmunol.169.5.2756. PMID 12193750
- [Background] Triebel F. LAG-3: a regulator of T-cell and DC responses and its use in therapeutic vaccination. Trends Immunol. 2003 Dec;24(12):619-22. doi: 10.1016/j.it.2003.10.001. PMID 14644131
- [Background] Buisson S, Triebel F. MHC class II engagement by its ligand LAG-3 (CD223) leads to a distinct pattern of chemokine and chemokine receptor expression by human dendritic cells. Vaccine. 2003 Feb 14;21(9-10):862-8. doi: 10.1016/s0264-410x(02)00533-9. PMID 12547595
- [Background] Andreae S, Buisson S, Triebel F. MHC class II signal transduction in human dendritic cells induced by a natural ligand, the LAG-3 protein (CD223). Blood. 2003 Sep 15;102(6):2130-7. doi: 10.1182/blood-2003-01-0273. Epub 2003 May 29. PMID 12775570
- [Background] El Mir S, Triebel F. A soluble lymphocyte activation gene-3 molecule used as a vaccine adjuvant elicits greater humoral and cellular immune responses to both particulate and soluble antigens. J Immunol. 2000 Jun 1;164(11):5583-9. doi: 10.4049/jimmunol.164.11.5583. PMID 10820232
- [Background] Prigent P, El Mir S, Dreano M, Triebel F. Lymphocyte activation gene-3 induces tumor regression and antitumor immune responses. Eur J Immunol. 1999 Dec;29(12):3867-76. doi: 10.1002/(SICI)1521-4141(199912)29:123.0.CO;2-E. PMID 10601994
- [Background] Cappello P, Triebel F, Iezzi M, Caorsi C, Quaglino E, Lollini PL, Amici A, Di Carlo E, Musiani P, Giovarelli M, Forni G. LAG-3 enables DNA vaccination to persistently prevent mammary carcinogenesis in HER-2/neu transgenic BALB/c mice. Cancer Res. 2003 May 15;63(10):2518-25. PMID 12750275
- [Background] Di Carlo E, Cappello P, Sorrentino C, D'Antuono T, Pellicciotta A, Giovarelli M, Forni G, Musiani P, Triebel F. Immunological mechanisms elicited at the tumour site by lymphocyte activation gene-3 (LAG-3) versus IL-12: sharing a common Th1 anti-tumour immune pathway. J Pathol. 2005 Jan;205(1):82-91. doi: 10.1002/path.1679. PMID 15586367
- [Background] Huard B, Tournier M, Hercend T, Triebel F, Faure F. Lymphocyte-activation gene 3/major histocompatibility complex class II interaction modulates the antigenic response of CD4+ T lymphocytes. Eur J Immunol. 1994 Dec;24(12):3216-21. doi: 10.1002/eji.1830241246. PMID 7805750
- [Background] Hannier S, Tournier M, Bismuth G, Triebel F. CD3/TCR complex-associated lymphocyte activation gene-3 molecules inhibit CD3/TCR signaling. J Immunol. 1998 Oct 15;161(8):4058-65. PMID 9780176
- [Background] Workman CJ, Vignali DA. The CD4-related molecule, LAG-3 (CD223), regulates the expansion of activated T cells. Eur J Immunol. 2003 Apr;33(4):970-9. doi: 10.1002/eji.200323382. PMID 12672063
- [Background] Macon-Lemaitre L, Triebel F. The negative regulatory function of the lymphocyte-activation gene-3 co-receptor (CD223) on human T cells. Immunology. 2005 Jun;115(2):170-8. doi: 10.1111/j.1365-2567.2005.02145.x. PMID 15885122
- [Background] Huang CT, Workman CJ, Flies D, Pan X, Marson AL, Zhou G, Hipkiss EL, Ravi S, Kowalski J, Levitsky HI, Powell JD, Pardoll DM, Drake CG, Vignali DA. Role of LAG-3 in regulatory T cells. Immunity. 2004 Oct;21(4):503-13. doi: 10.1016/j.immuni.2004.08.010. PMID 15485628
- [Background] Workman CJ, Vignali DA. Negative regulation of T cell homeostasis by lymphocyte activation gene-3 (CD223). J Immunol. 2005 Jan 15;174(2):688-95. doi: 10.4049/jimmunol.174.2.688. PMID 15634887
- [Background] Triebel F, Hacene K, Pichon MF. A soluble lymphocyte activation gene-3 (sLAG-3) protein as a prognostic factor in human breast cancer expressing estrogen or progesterone receptors. Cancer Lett. 2006 Apr 8;235(1):147-53. doi: 10.1016/j.canlet.2005.04.015. Epub 2005 Jun 8. PMID 15946792
- [Background] Lienhardt C, Azzurri A, Amedei A, Fielding K, Sillah J, Sow OY, Bah B, Benagiano M, Diallo A, Manetti R, Manneh K, Gustafson P, Bennett S, D'Elios MM, McAdam K, Del Prete G. Active tuberculosis in Africa is associated with reduced Th1 and increased Th2 activity in vivo. Eur J Immunol. 2002 Jun;32(6):1605-13. doi: 10.1002/1521-4141(200206)32:63.0.CO;2-6. PMID 12115643
- [Background] Immutep. 2006. ImmuFact IMP321 Product Information Brochure.
- [Background] Fougeray S, Brignone C, Triebel F. A soluble LAG-3 protein as an immunopotentiator for therapeutic vaccines: Preclinical evaluation of IMP321. Vaccine. 2006 Jun 29;24(26):5426-33. doi: 10.1016/j.vaccine.2006.03.050. Epub 2006 Mar 31. PMID 16621192
- [Background] Tseng JF, Willett CG, Fernandez-del Castillo C, Ryan DP, Clark JW, Zhu AX, Rattner DW, Winkelmann JL, Warshaw AL. Patients undergoing treatment for pancreatic adenocarcinoma can mount an effective immune response to vaccinations. Pancreatology. 2005;5(1):67-74. doi: 10.1159/000084492. Epub 2005 Mar 15. PMID 15775701
- [Background] Co, E.L.a., Gemcitabine Product Info. 2003.
- [Background] Series, M.H., 2003. MICROMEDEX, Greenwood Village, Colorado
- [Background] Hawkins WG, Gold JS, Dyall R, Wolchok JD, Hoos A, Bowne WB, Srinivasan R, Houghton AN, Lewis JJ. Immunization with DNA coding for gp100 results in CD4 T-cell independent antitumor immunity. Surgery. 2000 Aug;128(2):273-80. doi: 10.1067/msy.2000.107421. PMID 10923004
- [Background] Ko K, Yamazaki S, Nakamura K, Nishioka T, Hirota K, Yamaguchi T, Shimizu J, Nomura T, Chiba T, Sakaguchi S. Treatment of advanced tumors with agonistic anti-GITR mAb and its effects on tumor-infiltrating Foxp3+CD25+CD4+ regulatory T cells. J Exp Med. 2005 Oct 3;202(7):885-91. doi: 10.1084/jem.20050940. Epub 2005 Sep 26. PMID 16186187
- [Background] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu